CLINICAL TRIAL: NCT04046224
Title: A Phase I/II, Multicenter, Open-Label, Single-Dose, Dose-Ranging Study to Assess the Safety and Tolerability of ST-920, an AAV2/6 Human Alpha Galactosidase A Gene Therapy, in Subjects With Fabry Disease (STAAR)
Brief Title: Dose-Ranging Study of ST-920, an AAV2/6 Human Alpha Galactosidase A Gene Therapy in Subjects With Fabry Disease (STAAR)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST-920-201
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Fabry Disease
Keywords: Sangamo; Rare; Lysosomal Storage Disease; Gene Therapy
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequential dose escalation (Experimental): ST-920 is administered as a single infusion:
  1. Cohort 1: 0.5e13 vg/kg
  2. Cohort 2: 1.0e13 vg/kg
  3. Cohort 3: 3.0e13 vg/kg
  4. Cohort 4: 5.0e13 vg/kg
  Interventions: Biological: ST-920
- Expansion Cohorts (Experimental): 1. Anti Alpha-Gal A Antibody Positive Cohort
  2. Anti Alpha-Gal A Antibody Negative Cohort
  3. Female Cohort
  4. Renal Cohort
  5. Cardiac Cohort
  Interventions: Biological: ST-920

INTERVENTIONS:
Biological: ST-920 — Single dose of investigational product ST-920

SUMMARY:
This is the first in human treatment with ST-920, a recombinant AAV2/6 vector encoding the cDNA for human a-Gal A. The purpose of this study is to evaluate the safety and tolerability of ascending doses of ST-920. ST-920 aims to provide stable, long-term production of α-Gal A at therapeutic levels in subjects with Fabry disease. The constant production of α-Gal A in humans should, importantly, enable reduction and potentially clearance of Fabry disease substrates Gb3 and lyso-Gb3. On Day 1, patients will be infused intravenously with a single dose of ST-920 and followed for a period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Documented diagnosis of Fabry disease
* One or more of the following symptoms: i) cornea verticillata, ii) acroparesthesia, iii) anhidrosis, iv) angiokeratoma
* Subject must be fully vaccinated (as per the Centers for Disease Control and Prevention (CDC) definition in the US and as per local guidelines in other countries) for COVID-19 at least one month prior to dosing

Additional Inclusion Criteria:

Renal Cohort:

* Screening eGFR value between 40-90 mL/min/1.73 m²
* Linear negative eGFR slope (estimated from at least 3 serum creatinine values within 18 months, including the value obtained during screening visit) of ≥ 2 mL/min/1.73m²/year

Cardiac Cohort:

• Left ventricular hypertrophy (LVH) in 2D echocardiography or CMR defined as an end diastolic septum and posterior wall thickness ≥12 mm with no other explanation for LVH, OR presentation with cardiac changes indicative of disease progression such as decreased global longitudinal strain on 2D strain echocardiography or low native T1 mapping on CMR

Exclusion Criteria:

* Neutralizing antibodies to AAV6
* eGFR < 40 ml/min/1.73m2
* New York Heart Association Class III or higher
* Active infection with hepatitis A, B or C, HIV or TB
* History of liver disease such as clinically significant steatosis, fibrosis, non-alcoholic steatohepatitis (NASH) and cirrhosis, biliary disease within 6 months of informed consent; except for Gilbert's syndrome
* Elevated circulating serum AFP
* Recent or recurrent hypersensitivity response to ERT within within 6 months prior to consent
* Current or history of systemic (IV or oral) immunomodulatory agents, or biologics or steroid use in the past 6 months prior to consent (topical treatment and inhaled allowed).
* Contraindication to use of corticosteroids
* History of malignancy except for non-melanoma skin cancer and localized prostate cancer treated with curative intent
* Recent history of alcohol or substance abuse
* Participation in investigational interventional drug or medical device study throughout the duration of this study and within previous 3 months prior to consent
* Prior treatment with a gene therapy product
* Known hypersensitivity to components of ST-920 formulation
* Any other reason that, in the opinion of the Site Investigator or Medical Monitor, would render the subject unsuitable for participation in the study including but not limited to risk of COVID-19 infection

Additional exclusion criteria for:

Renal cohort:

* History of renal dialysis or transplantation
* History of acute kidney insufficiency in the 6 months prior to screening
* Angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) therapy initiated within 4 weeks prior to screening or changed ACE inhibitor or ARB dose in the 4 weeks prior to screening
* Urine protein to creatinine ratio (UPCR) > 0.5 g/g who are not being treated with an ACE inhibitor or ARB

Cardiac cohort:

* Significant cardiac fibrosis defined by late gadolinium enhancement on CMR
* Any contraindications to CMR as per local hospital/institution guidelines
* Angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) therapy initiated within 4 weeks prior to screening or changed ACE inhibitor or ARB dose in the 4 weeks prior to screening
* NYHA Class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 12 months after the ST-920 infusion
  Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) in subjects who receive ST-920 as assessed by Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics, Inc.
Locations (18):
- United States (9):
  - University of California, Irvine, Irvine, California
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mt. Sinai School of Medicine, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Lysosomal and Rare Disorders Research and Treatment Center (LDRTC), Fairfax, Virginia
- The Royal Melbourne Hospital, Parkville, Victoria, Australia
- M.A.G.I.C. Clinic Ltd., Calgary, Alberta, Canada
- Germany (2):
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - University Hospital of Würzburg, Würzburg
- Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany, Italy
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Royal Free Hospital, London